CLINICAL TRIAL: NCT01323374
Title: A Phase II, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Dose-Response, Study To Assess The Clinical Benefit Of Droxidopa and Droxidopa/Carbidopa In Subjects With Fibromyalgia
Brief Title: Study To Assess The Clinical Benefit Of Droxidopa And Droxidopa/Carbidopa In Subjects With Fibromyalgia
Acronym: FMS201
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chelsea Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Droxidopa FMS201
Record Dates: First submitted 2011-03-24; First posted 2011-03-25 (Estimated); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; FMS; droxidopa; pain
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — Droxidopa; 3,4-dihydroxyphenylserine aldolase; Carbidopa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (12):
- Droxidopa 200mg TID (Experimental)
  Interventions: Drug: Droxidopa
- Droxidopa 400mg TID (Experimental)
  Interventions: Drug: Droxidopa
- Droxidopa 600mg TID (Experimental)
  Interventions: Drug: Droxidopa
- Carbidopa 25mg TID (Active Comparator)
  Interventions: Drug: Carbidopa
- Carbidopa 50 mg TID (Active Comparator)
  Interventions: Drug: Carbidopa
- Droxidopa/carbidopa 200mg/25mg TID (Experimental)
  Interventions: Drug: Droxidopa/carbidopa
- Droxidopa/carbidopa 400mg/25mg TID (Experimental)
  Interventions: Drug: Droxidopa/carbidopa
- Droxidopa/carbidopa 600mg/25mg TID (Experimental)
  Interventions: Drug: Droxidopa/carbidopa
- Droxidopa/carbidopa 200mg/50mg TID (Experimental)
  Interventions: Drug: Droxidopa/carbidopa
- Droxidopa/carbidopa 400mg/50mg TID (Experimental)
  Interventions: Drug: Droxidopa/carbidopa
- Droxidopa/carbidopa 600mg/50mg TID (Experimental)
  Interventions: Drug: Droxidopa/carbidopa
- Placebo TID (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Droxidopa — Oral, 200mg, 400mg or 600mg TID, duration includes up to a 1 week blinded titration period followed by an 8 week treatment period.
  Other Names: L-threo-3,4-dihydroxyphenylserine; L-threo-DOPS; L-DOPS
  Arms: Droxidopa 200mg TID; Droxidopa 400mg TID; Droxidopa 600mg TID
Drug: Carbidopa — Oral, 25mg, or 50mg TID, duration includes up to a 1 week blinded titration period followed by an 8 week treatment period.
  Other Names: Lodosyn
  Arms: Carbidopa 25mg TID; Carbidopa 50 mg TID
Drug: Droxidopa/carbidopa — Oral, 200mg/25mg, 400mg/25mg, 600mg/25mg, 200mg/50mg, 400mg/50mg, or 600mg/50mg TID. Duration includes up to a 1 week titration period followed by an 8 week treatment period.
  Other Names: L-threo-3,4-dihydroxyphenylserine / Lodosyn; L-threo-DOPS / Lodosyn; L-DOPS / Lodosyn
  Arms: Droxidopa/carbidopa 200mg/25mg TID; Droxidopa/carbidopa 200mg/50mg TID; Droxidopa/carbidopa 400mg/25mg TID; Droxidopa/carbidopa 400mg/50mg TID; Droxidopa/carbidopa 600mg/25mg TID; Droxidopa/carbidopa 600mg/50mg TID
Drug: Placebo — Oral, placebo TID
  Other Names: Inactive ingrediant
  Arms: Placebo TID

SUMMARY:
A correlation between increased norepinephrine concentration in the central nervous system (CNS) and a decrease in fibromyalgia pain has been suggested in clinical studies. Therefore, as a pro-drug of norepinephrine, droxidopa could potentially benefit fibromyalgia patients by reducing pain as a result of increasing CNS levels of norepinephrine.

As this benefit is presumed to be a central effect, the addition of carbidopa, a peripheral DOPA decarboxylase (DDC) inhibitor, may favorably impact the drug's treatment profile. Carbidopa is utilized as a blocker of peripheral DDC, an enzyme required for the conversion of droxidopa into norepinephrine. Therefore, inhibition of peripheral DDC should result in a reduction of any side effects resulting from the peripheral production of norepinephrine, whilst allowing for increased central levels, and hence, increased centrally mediated benefits.

The purpose of the study is the obtain information regarding the proper dosing, effectiveness and safety of droxidopa and combination droxidopa/carbidopa treatments in patients with fibromyalgia.

DETAILED DESCRIPTION:
Fibromyalgia syndrome (FMS) and Chronic widespread pain (CWP) are two syndromes within a broader class known as functional somatic syndromes. Chronic widespread pain (CWP) is defined according to the American College of Rheumatology (ACR), as pain both above and below the waist involving both sides of the body and lasting for at least 3 months. Fibromyalgia syndrome (FMS), a subset of CWP, is a multisystem disease characterized by sleep disturbance, fatigue, headache, morning stiffness, paresthesias, and anxiety.

While there is debate as to specific etiology and pathogenesis, fibromyalgia is generally believed to be the result of a perturbation of central pain processing, specifically the neuroendocrine system. Fibromyalgia patients have been shown to have lower levels of metabolites from three neurotransmitters (serotonin, norepinephrine, and dopamine) in their cerebrospinal fluid (CSF) compared to healthy controls. The low rate of turnover of these neurotransmitters supports the hypothesis of a metabolic defect in fibromyalgia and suggests that the defect occurs at a neuroregulatory level. Results of a study that examined the effect of a permanent reduction in the noradrenergic innervation of the spinal cord suggested that the antinociceptive effects of norepinephrine are closely linked to opioidergic and tachykinergic neurotransmission.

Droxidopa [also, known as L-threo-3,4-dihydroxyphenylserine, L-threo-DOPS, or L-DOPS] is the International non-proprietary name (INN) for a synthetic amino acid precursor of norepinephrine (NE), which was originally developed by Sumitomo Pharmaceuticals Co., Limited, Japan. It has been approved for use in Japan since 1989. Droxidopa has been shown to improve symptoms of orthostatic hypotension that result from a variety of conditions including Shy Drager syndrome (Multiple System Atrophy), Pure Autonomic Failure, and Parkinson's disease. There are four stereoisomers of DOPS; however, only the L-threo-enantiomer (droxidopa) is biologically active. Data from clinical studies and post-marketing surveillance programs conducted in Japan show that the most commonly reported adverse drug reactions with droxidopa are increased blood pressure, nausea, and headache. In clinical studies to date, data suggests that droxidopa is well-tolerated and effective as a norepinephrine precursor.

Pre-clinical and clinical studies suggest that droxidopa has an analgesic effect in patients with chronic pain. An increase in central nervous system (CNS) levels of norepinephrine has been shown to correlate with an analgesic effect. Based on the pre-clinical and clinical findings to date, it is hypothesized that droxidopa can provide pain reduction in fibromyalgia patients through increasing the CNS levels of norepinephrine.

Carbidopa is a DOPA decarboxylase (DDC) inhibitor. At therapeutic doses carbidopa does not cross the blood-brain barrier and therefore should not inhibit CNS metabolism of droxidopa to NE. Decreasing the activity of DDC in the periphery enables droxidopa metabolism to be focused in the CNS. This CNS focus should increase CNS response while also limiting the increase in blood pressure associated with peripheral droxidopa metabolism. In addition, as DDC is an enzyme required for the conversion of droxidopa into its active metabolite norepinephrine, inhibition of peripheral DDC, utilizing Carbidopa, should result in a reduction of any side effects resulting from the peripheral production of NE, whilst allowing for increased central levels, and hence, increased centrally mediated benefits.

The primary objective of this study is to determine the efficacy of droxidopa and droxidopa/carbidopa in the treatment of pain associated with fibromyalgia. Secondary objectives include: evaluation of the effect of droxidopa and combinations of droxidopa/carbidopa on signs and symptoms of fibromyalgia, evaluation of the effect of droxidopa and combinations of droxidopa/carbidopa on the overall quality of life of fibromyalgia patients, evaluation of the dose-response relationship for droxidopa between different doses of droxidopa, carbidopa and combinations of droxidopa/carbidopa in fibromyalgia patients, evaluation of the clinical benefit of treatment with different doses of droxidopa, carbidopa and combinations of droxidopa/carbidopa in fibromyalgia patients, estimation of the optimal dose for relief of fibromyalgia pain using response surface methodology, and evaluation of the safety of droxidopa and droxidopa/carbidopa treatments.

ELIGIBILITY:
Inclusion Criteria:

* Male or female and aged 18 years or over
* Clinical diagnosis of fibromyalgia as defined by the 1990 American College of Rheumatology (ACR) criteria
* Provide written informed consent to participate in the study and understand that they may withdraw their consent at any time without prejudice to their future medical care
* Have a score of between 20mm and 90mm on the Visual Analog Scale for Pain (VAS-P) section of the SF-MPQ at screening and baseline visits

Exclusion Criteria:

* Have uncontrolled hypertension (defined as systolic blood pressure >160 mmHg and/or diastolic blood pressure >110 mmHg) or use of ≥2 antihypertensive medications
* Patients currently taking pregabalin; unless they provide written informed consent and agree to discontinue pregabalin use 3 weeks prior to other screening procedures and for the duration of the study
* Currently taking tri-cyclic antidepressant medication
* Currently taking any norepinephrine re-uptake inhibitors
* Have clinically relevant depression noted as significant by a score greater than 17 on the Hamilton Depression Scale (HAM-D)
* History of known or suspected drug or substance abuse
* Women of childbearing potential who are not using a medically accepted contraception (Reproductive potential: Female subjects should be either post-menopausal (amenorrhea for at least 12 consecutive months), surgically sterile, or women of child-bearing potential (WOCP) who are using or agree to use acceptable methods of contraception throughout the study period and for 4 weeks after the last dose of investigational product. Acceptable contraceptives include intrauterine devices (IUDs), hormonal contraceptives (oral, depot, patch or injectable) and double barrier methods such as condoms or diaphragms with spermicidal gel or foam. If hormonal contraceptives are used they should be taken according to the package insert. WOCP who are not currently sexually active must agree to use acceptable contraception, as defined above, if they decide to become sexually active during the period of the study and for 4 weeks after the last dose of investigational product. For WOCP a urine pregnancy test must be conducted at screening, baseline and study termination; the results must be negative at screening and at baseline. Any positive result will be confirmed by serum beta HCG pregnancy test).
* Sexually active males whose partner is a WOCP must agree to use condoms for the duration of the study and for 4 weeks after the last dose
* Women who are pregnant, breast feeding, or plan to become pregnant during the course of this study
* Known or suspected hypersensitivity to the study medication or any of its ingredients
* Have in the investigator's opinion any significant cardiac arrhythmia
* Any significant systemic, hepatic, cardiac or renal illness
* Diabetes mellitus or insipidus
* Have a history of closed angle glaucoma
* Have a known or suspected current malignancy. Patients with a history of cancer must be symptom- and treatment-free for at least 5 years prior to randomization, with the exception of patients with non-melanoma, non-invasive skin cancers (such as basal cell carcinoma), who should not have had an intervention or recurrence within one year of starting the study
* Patients with known gastrointestinal illness or other gastrointestinal disorder that may, in the investigator's opinion, affect the absorption of study drug
* In the investigator's opinion, have clinically significant abnormalities on clinical examination or laboratory testing
* In the investigator's opinion, are unable to adequately co-operate because of individual or family situation
* In the investigator's opinion, are suffering from a mental disorder that interferes with the diagnosis and/or with the conduct of the study, e.g. schizophrenia, major depression, dementia
* Are not able or willing to comply with the study requirements for the duration of the study
* Have participated in another clinical trial with an investigational agent (including named patient or compassionate use protocol) within 1 month before the start of the study
* Previous enrollment in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2009-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Determine the efficacy of droxidopa and droxidopa/carbidopa in the treatment of pain associated with fibromyalgia | Baseline to end of 8 week treatment period

SECONDARY OUTCOMES:
Evaluate the effect of droxidopa and combinations of droxidopa/carbidopa on signs and symptoms of fibromyalgia (including depression, fatigue, and sleep disorder) | Baseline to end of 8 week treatment period
Evaluate the effect of droxidopa and combinations of droxidopa/carbidopa on the overall quality of life of fibromyalgia patients | Baseline to end of 8 week treatment period
Evaluate the dose-response relationship for droxidopa (200, 400, and 600mg TID), carbidopa (25 and 50mg TID) and combinations of droxidopa/carbidopa (200/25, 200/50, 400/25, 400/50, 600/25 and 600/50mg TID) in the treatment of fibromyalgia patients | Baseline to end of 8 week treatment period
Evaluate the clinical benefit of treatment with 200, 400, and 600mg droxidopa TID, or 25 and 50mg carbidopa TID and combinations of droxidopa/carbidopa 200/25, 200/50, 400/25, 400/50, 600/25 and 600/50mg TID in the treatment of fibromyalgia patients | Baseline to end of 8 week treatment period
Estimate the optimal dose for relief of fibromyalgia pain using response surface methodology | Baseline to end of 8 week treatment period
Evaluate the safety of droxidopa and droxidopa/carbidopa treatments based on the occurrence of treatment-emergent adverse events (AE) and specific evaluation of blood pressure, heart rate, ECG, and laboratory findings across the study. | Baseline to end of 4 week follow-up period following 8 week treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Ernest Choy, M.D., Principal Investigator — Academic Dept of Rheumatology Kings College London
Locations (7):
- United Kingdom (7):
  - Rheumatology Department; Barnsley Hospital NHS Foundation Trust, Barnsley
  - MAC UK Neuroscience, Liverpool
  - Academic Dept of Rheumatology, Kings College London, London
  - MAC UK Neuroscience, Manchester
  - Musculoskeletal Department; Freeman Hospital, Newcastle upon Tyne
  - Rheumatology Department, Poole Hospital NHS Trust, Poole
  - Clinical Trials Unit; Main Hospital; Salford Rooyal NHS Foundation Trust, Salford

REFERENCES:
- See also: EudraCT summary results — https://www.clinicaltrialsregister.eu/ctr-search/trial/2008-001123-62/results